CLINICAL TRIAL: NCT00795691
Title: High and Low Carbohydrate Weight Loss Approaches to Type 2 Diabetes Mellitus (The Diabetes Dietary Study (DDS))
Brief Title: Diabetes Dietary Study- Low Carbohydrate and Low-Fat Diets in Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: Robert C. Atkins Foundation (Other)
Responsible Party: Principal Investigator, Judith Wylie-Rosett, Professor, Department of Epidemiology and Population Health, Albert Einstein College of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2002-180
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Type 2 Diabetes
Keywords: diabetes; low-carbohydrate diet; weight loss; obesity; dietary intervention
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus; Weight Loss; Obesity | interventions — Diet, Carbohydrate-Restricted; Diet, Fat-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Low-carbohydrate diet (Experimental): The low-carbohydrate diet was based on the Atkins weight loss diet. The daily intake goals were to restrict intake of carbohydrate to 20-25 grams for the first 2-week phase. If body weight decreased, the daily goal for carbohydrate was increased by 5 grams. If body weight increased, the daily goal for carbohydrate intake was decreased by 5 grams. The minimum goal for carbohydrate intake was 20 grams per day and the maximum goal was 50 grams per day.
  Interventions: Behavioral: low-carbohydrate diet
- Low-fat diet (Active Comparator): The low-fat diet was based on the algorithm used to restrict fat and calorie intake in the Diabetes Prevention Program. The daily goals for fat intake was based on an algorithm to reduce total calorie intake to achieve a one pound weight loss per week with 25% of calories from fat.
  Interventions: Behavioral: low-fat diet

INTERVENTIONS:
Behavioral: low-carbohydrate diet — ketogenic low-carbohydrate diet in patients with type 2 diabetes
  Arms: Low-carbohydrate diet
Behavioral: low-fat diet — low-fat diet in patients with type 2 diabetes
  Arms: Low-fat diet

SUMMARY:
The purpose of this study is to determine the effects of a low-carbohydrate diet compared to a low-fat/high-carbohydrate diet on glucose control in patients who have Type 2 Diabetes.

DETAILED DESCRIPTION:
Obesity is not only a risk factor for type 2 diabetes but it also frequently increases the need for insulin requirement in people with type 2 diabetes who are overweight or obese. However, since insulin is a lipogenic hormone, insulin or sulfonylurea therapy that increases circulating insulin levels often results in additional weight gain. Controlled-carbohydrate "ketogenic" diets have been popular as an alternative way of losing weight, but little is known about the safety and efficacy of using a ketogenic approach in the management of overweight/obese patients with type 2 diabetes.

The proposed study will randomize a group of 126 overweight or obese (BMI > 25 and < 40) adults with type 2 diabetes to either a low-carbohydrate or a low-fat weight loss diet. The primary study endpoint will be six and twelve month changes in glycemic control as measured by hemoglobin A1c (HbA1c). Secondary endpoints include adiposity (BMI, body composition and fat distribution); blood glucose patterns (from self-monitoring records); change in antidiabetic medications (potential decrease in number and dosage), lipids, insulin sensitivity from a meal tolerance test, other metabolic markers (C-reactive protein, leptin) and participants' lifestyle (physical activity and diet) and perceptions of satiety, quality of life, mood, and well-being.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 2 diabetes
* HbA1c 7-10%
* BMI (kg/m2) > 25 and < 40 and weight < 280 lb.
* Skill at and willingness to perform capillary blood glucose self-monitoring ---Insulin (changed to long-acting basal during run-in) or sulfonylurea treatment

Exclusion Criteria:

* Age > 65
* Weight >280 lb
* Health conditions that may interfere with study participation or for which the study interventions may be contraindicated. These include: kidney stones or kidney disease (creatinine > 1.3 and 1.5 mg/dL for females and males, respectively; proteinuria > 300 ug/g creatinine); liver or gall bladder disease; significant heart disease (myocardial infarction in the past six months, prior or current evidence of congestive heart failure, other evidence of left ventricular (LV) dysfunction) or other indices of active cardiac abnormalities, (angina, electrocardiogram evidence of ischemia or transmural myocardial infarction), significant anemia; and cancer (other than effectively treated non melanomatous skin cancer and surgically treated cervical cancer in situ).
* Current hypokalemia defined as serum potassium levels <3.5 mg/dL.
* Osteoporosis
* Type 1 diabetes (history of ketoacidosis or undetectable fasting C-peptide levels)
* History of severe or repeated hypoglycemia, or hypoglycemia unawareness. Lack of recourse to another person in the immediate vicinity in the unlikely event that they require outside assistance for severe hypoglycemia.
* Triglyceride levels > 400 mg/dL.
* Inability or unwillingness to comply with any aspects of the dietary and research protocol.
* Weight changes > 10 lbs in the past three months.
* History of binge eating disorder or other eating disorders.
* Pregnancy or intention to become pregnant in the next 12 months.
* Current oral hypoglycemic medication that raises the blood insulin level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2004-05; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c at month 3 | 3 months into treatment
  Hemoglobin A1c (HbA1c) is a form of hemoglobin (a blood pigment that carries oxygen) that is bound to glucose. HbA1c level indicates blood glucose levels over the previous 2 - 3 months. HbA1c values between 4 and 5.6 are considered normal. HbA1c values greater than 6.5 indicate diabetes.
Hemoglobin A1c at month 6 | 6 months into treatment
  Hemoglobin A1c (HbA1c) is a form of hemoglobin (a blood pigment that carries oxygen) that is bound to glucose. HbA1c level indicates blood glucose levels over the previous 2 - 3 months. HbA1c values between 4 and 5.6 are considered normal. HbA1c values greater than 6.5 indicate diabetes.
Hemoglobin A1c at month 12 | 12 months into treatment
  Hemoglobin A1c (HbA1c) is a form of hemoglobin (a blood pigment that carries oxygen) that is bound to glucose. HbA1c level indicates blood glucose levels over the previous 2 - 3 months. HbA1c values between 4 and 5.6 are considered normal. HbA1c values greater than 6.5 indicate diabetes.
Change in Body Weight at month 3 | Baseline and 3 months into treatment
  Change in body weight often reflects the effects of dietary changes. Generally, an increase in body weight is correlated with increasing blood glucose levels while a decrease in body weight correlates to decreasing blood glucose levels. Dietary changes that result in decreased body weight will be associated with better glucose control.
Change in Body Weight at month 6 | Baseline and 6 months into treatment
  Change in body weight often reflects the effects of dietary changes. Generally, an increase in body weight is correlated with increasing blood glucose levels while a decrease in body weight correlates to decreasing blood glucose levels. Dietary changes that result in decreased body weight will be associated with better glucose control.
Change in Body Weight at month 12 | Baseline and 12 months into treatment
  Change in body weight often reflects the effects of dietary changes. Generally, an increase in body weight is correlated with increasing blood glucose levels while a decrease in body weight correlates to decreasing blood glucose levels. Dietary changes that result in decreased body weight will be associated with better glucose control.

SECONDARY OUTCOMES:
Change in Body Fat at month 6 | Baseline and 6 months into treatment
  A bioelectrical impedance analysis scale is used to measure body fat. Having a higher proportion of body fat is associated with poorer blood glucose control.
Change in Body Fat at month 12 | Baseline and 12 months into treatment
  A bioelectrical impedance analysis scale is used to measure body fat. Having a higher proportion of body fat is associated with poorer blood glucose control.
Change in Lean Body Mass at month 6 | Baseline and 6 months into treatment
  A bioelectrical impedance analysis scale is used to measure lean body mass. Having a higher proportion of lean body mass is associated with better blood sugar control.
Change in Lean Body Mass at month 12 | Baseline and 12 months into treatment
  A bioelectrical impedance analysis scale is used to measure lean body mass. A higher proportion of lean mass is associated with better blood sugar control.
Change in antidiabetic medication dosage at month 3 | Baseline and 3 months into treatment
  If medication dosage is reduced, it generally indicates that blood glucose is better controlled. If dosage increases, it generally indicates that blood glucose was not well controlled.
Change in antidiabetic medication dosage at month 6 | Baseline and 6 months into treatment
  If medication dosage is reduced, it generally indicates that blood glucose is better controlled. If dosage increases, it generally indicates that blood glucose was not well controlled.
Change in antidiabetic medication dosage at month 12 | Baseline and 12 months into treatment
  If medication dosage is reduced, it generally indicates that blood glucose is better controlled. If dosage increases, it generally indicates that blood glucose was not well controlled.
Change in insulin sensitivity at month 6 | Baseline and 6 months into treatment
  Insulin sensitivity is calculated from the fasting blood glucose and insulin levels derived from laboratory tests. An increase in insulin sensitivity relates to better blood glucose control. A reduction in insulin sensitivity is related to poorer blood glucose control.
Total Cholesterol at month 6 | 6 months into treatment
  Blood level of total cholesterol measures cardiovascular risk. Total cholesterol is reduced with weight loss. The change would be an indication of reduction in cardiovascular risk.
Total Cholesterol at month 12 | 12 months into treatment
  Blood level of total cholesterol measures cardiovascular risk. Total cholesterol is reduced with weight loss. The change would be an indication of reduction in cardiovascular risk.
High-density lipoprotein cholesterol at month 6 | 6 months into treatment
  Blood level of high density lipoprotein (HDL) cholesterol, measures cardiovascular risk. HDL cholesterol is expected to increase with weight loss. The change would be an indication of reduction in cardiovascular risk.
High-density lipoprotein cholesterol at month 12 | 12 months into treatment
  Blood level of high density lipoprotein (HDL) cholesterol, measures cardiovascular risk. HDL cholesterol is expected to increase with weight loss. The change would be an indication of reduction in cardiovascular risk.
Low-density lipoprotein cholesterol at month 6 | 6 months into treatment
  Low density lipoproteins (LDL) cholesterol measures cardiovascular risk. LDL cholesterol is expected to be reduced with weight loss. This change would be an indication of reduction in cardiovascular risk.
Low-density lipoprotein cholesterol at month 12 | 12 months into treatment
  Low density lipoprotein (LDL) cholesterol measures cardiovascular risk. LDL cholesterol is expected to be reduced with weight loss. This change would be an indication of reduction in cardiovascular risk.
Triglycerides at month 6 | 6 months into treatment
  Blood Triglyceride levels measure cardiovascular risk. Triglycerides are expected to be reduced with weight loss. This change would be an indication of reduction in cardiovascular risk.
Triglycerides cholesterol at month 12 | 12 months into treatment
  The blood level of triglycerides measures cardiovascular risk. Triglycerides are expected to be reduced with weight loss. This change would be an indication of reduction in cardiovascular risk.
Dietary caloric intake as assessed using the Dietary History Questionnaire (DHQ) at month 6 | 6 months into treatment
  Dietary intake is assessed using the Dietary History Questionnaire (DHQ), a web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total energy (calories) consumed are based on the nutrient values from NHANES. It is anticipated that a decrease in calorie intake would result in body weight reduction which normally correlates to increased blood glucose control. Likewise, an increase in calories generally result in body weight increase which correlates to decreased blood glucose control.
Dietary caloric intake as assessed using the Dietary History Questionnaire (DHQ) at month 12 | 12 months into treatment
  Dietary intake is assessed using the Dietary History Questionnaire (DHQ), a web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total energy (calories) consumed are based on the nutrient values from NHANES. It is anticipated that a decrease in calorie intake would result in body weight reduction which normally correlates to increased blood glucose control. Likewise, an increase in calories generally result in body weight increase which correlates to decreased blood glucose control.
Dietary carbohydrate intake as assessed using the Dietary History Questionnaire (DHQ) at month 6 | 6 months into treatment
  Dietary carbohydrate intake is assessed using the Dietary History Questionnaire (DHQ), which is web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total intake (in grams) of carbohydrates are based on the nutrient values from NHANES. It is anticipated that an increase in carbohydrate intake would result in an increase in blood HbA1c level, and a decrease in carbohydrate intake would result in a decrease in the blood HbA1c level.
Dietary carbohydrate intake as assessed using the Dietary History Questionnaire (DHQ) at month 12 | 12 months into treatment
  Dietary carbohydrate intake is assessed using the Dietary History Questionnaire (DHQ), which is web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total intake (in grams) of carbohydrates are based on the nutrient values from NHANES. It is anticipated that an increase in carbohydrate intake would result in an increase in blood HbA1c level, and a decrease in carbohydrate intake would result in a decrease in the blood HbA1c level.
Dietary fat intake as assessed using the Dietary History Questionnaire (DHQ) at month 6 | 6 months into treatment
  Dietary fat intake is assessed using the Dietary History Questionnaire (DHQ), which is web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total intake (in grams) of fat (saturated fat, monounsaturated fat and polyunsaturated fat) are based on the nutrient values from NHANES. It is anticipated that an increase in fat intake would result in an increase in total and LDL blood cholesterol levels, and a decrease in fat intake would result in a decrease in total and LDL blood cholesterol levels.
Dietary fat intake as assessed using the Dietary History Questionnaire (DHQ) at month 12 | 12 months into treatment
  Dietary fat intake is assessed using the Dietary History Questionnaire (DHQ), which is web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total intake (in grams) of fat (saturated fat, monounsaturated fat and polyunsaturated fat) are based on the nutrient values from NHANES. It is anticipated that an increase in fat intake would result in an increase in total and LDL blood cholesterol levels, and a decrease in fat intake would result in a decrease in total and LDL blood cholesterol levels.
Dietary protein intake as assessed using the Dietary History Questionnaire (DHQ) at month 6 | 6 months into treatment
  Dietary protein intake is assessed using the Dietary History Questionnaire (DHQ), which is web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total intake (in grams) of protein are based on the nutrient values from NHANES. It is anticipated that an increase in protein intake (relative to carbohydrate) will result in loss of body fat and reduction in body weight, while a decrease in protein intake(relative to carbohydrate) will result in increased body fat and body weight.
Dietary protein intake as assessed using the Dietary History Questionnaire (DHQ) at month 12 | 12 months into treatment
  Dietary protein intake is assessed using the Dietary History Questionnaire (DHQ), which is web-based food frequency questionnaire. Participants select the serving size and frequency of intake for the foods listed. The items listed and serving size choices are derived from the National Health and Nutrition Examination Survey (NHANES). Calculations of total intake (in grams) of protein are based on the nutrient values from NHANES. It is anticipated that an increase in protein intake (relative to carbohydrate) will result in loss of body fat and reduction in body weight, while a decrease in protein intake(relative to carbohydrate) will result in increased body fat and body weight.
Physical activity was assessed by patient self-report at month 6 | 6 months into treatment
  Physical activity was assessed using the Modifiable Physical activity Questionnaire (MAQ) with the 7-Day Physical Activity Recall interview. Participants were asked to provide information about the frequency, duration and intensity of various physical activities. MAQ responses and 7-day recall data were coded and entered into software program, which was designed to calculate average daily energy expenditure. Participants were instructed to avoid changing physical activity while in the study because change in physical activity could confound assessment of the dietary questions. An increase in physical activity could increase loss of body weight and reduction in blood HbA1c. A decrease in physical activity could increase body weight and increase HbA1c.
Physical activity was assessed by patient self-report at month 12 | 12 months into treatment
  Physical activity was assessed using the Modifiable Physical activity Questionnaire (MAQ) with the 7-Day Physical Activity Recall interview. Participants were asked to provide information about the frequency, duration and intensity of various physical activities. MAQ responses and 7-day recall data were coded and entered into software program, which was designed to calculate average daily energy expenditure. Participants were instructed to avoid changing physical activity while in the study because change in physical activity could confound assessment of the dietary questions. An increase in physical activity could increase loss of body weight and reduction in blood HbA1c. A decrease in physical activity could increase body weight and increase HbA1c.
Quality of life as assessed using the Diabetes Quality of Life Scale at month 6 | 6 months into treatment
  Quality of Life is assessed using the Diabetes Quality of Life (DQOL) questionnaire. The DQOL questionnaire contains 62 items which participants rank from 1(very satisfied) to 5 (very dissatisfied). The score gives an indication of participants' satisfaction with treatment in terms of level of well-being and disability. The total score ranges from 0 to 310. The score is negatively correlated to Quality of Life with higher scores indicating higher dissatisfaction and therefore, lower perceived Quality of Life. It is expected that reduction in the blood HbA1c level will be associated with an increase in the Diabetes Quality of Life (i.e. a decrease in DQOL score), and an increase in the HbA1c level will correlate to a lower Diabetes Quality of Life (i.e. an increase in DQOL score).
Quality of life as assessed using the Diabetes Quality of Life Scale at month 12 | 12 months into treatment
  Quality of Life is assessed using the Diabetes Quality of Life (DQOL) questionnaire. The DQOL questionnaire contains 62 items which participants rank from 1(very satisfied) to 5 (very dissatisfied). The score gives an indication of participants' satisfaction with treatment in terms of level of well-being and disability. The total score ranges from 0 to 310. The score is negatively correlated to Quality of Life with higher scores indicating higher dissatisfaction and therefore, lower perceived Quality of Life. It is expected that reduction in the blood HbA1c level will be associated with an increase in the Diabetes Quality of Life (i.e. a decrease in DQOL score), and an increase in the HbA1c level will correlate to a lower Diabetes Quality of Life (i.e. an increase in DQOL score).

CONTACTS AND LOCATIONS:
Overall Officials: Judith Wylie-Rosett, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Albert Einstein College of Medicine, General Clinical Research Center, The Bronx, New York, United States

REFERENCES:
- [Background] Cunningham C, Johnson S, Cowell B, Soroudi N, Segal-Isaacson CJ, Davis NJ, Isasi CR, Wylie-Rosett J. Menu plans in a diabetes self-management weight loss program. J Nutr Educ Behav. 2006 Jul-Aug;38(4):264-6. doi: 10.1016/j.jneb.2006.01.013. No abstract available. PMID 16785099
- [Background] Davis NJ, Cohen HW, Wylie-Rosett J, Stein D. Serum potassium changes with initiating low-carbohydrate compared to a low-fat weight loss diet in type 2 diabetes. South Med J. 2008 Jan;101(1):46-9. doi: 10.1097/SMJ.0b013e31815d2696. PMID 18176291
- [Result] Davis NJ, Tomuta N, Schechter C, Isasi CR, Segal-Isaacson CJ, Stein D, Zonszein J, Wylie-Rosett J. Comparative study of the effects of a 1-year dietary intervention of a low-carbohydrate diet versus a low-fat diet on weight and glycemic control in type 2 diabetes. Diabetes Care. 2009 Jul;32(7):1147-52. doi: 10.2337/dc08-2108. Epub 2009 Apr 14. PMID 19366978
- [Derived] Davis NJ, Tomuta N, Isasi CR, Leung V, Wylie-Rosett J. Diabetes-specific quality of life after a low-carbohydrate and low-fat dietary intervention. Diabetes Educ. 2012 Mar-Apr;38(2):250-5. doi: 10.1177/0145721711436132. Epub 2012 Feb 7. PMID 22316641
- [Derived] Davis NJ, Crandall JP, Gajavelli S, Berman JW, Tomuta N, Wylie-Rosett J, Katz SD. Differential effects of low-carbohydrate and low-fat diets on inflammation and endothelial function in diabetes. J Diabetes Complications. 2011 Nov-Dec;25(6):371-6. doi: 10.1016/j.jdiacomp.2011.08.001. Epub 2011 Oct 27. PMID 22036100